CLINICAL TRIAL: NCT03737058
Title: Joint Oncology Collaboration for Proactive Symptom Assessments by a Lay Health Worker
Brief Title: Lay Health Worker Led Symptom Assessment Intervention
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor, Stanford University
Other Study IDs: SU12
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Program participants — The intervention is a 12-month telephonic program in which a lay health worker (LHW), supervised on-site by a registered nurse practitioner (RNP), assessed patient symptoms after diagnosis using the validated Edmonton Symptom Assessment Scale (ESAS) (cite) with the frequency of symptom assessment varying based on patient risk.

SUMMARY:
Rising costs and poor patient experiences from under-treated symptoms have led to the demand for approaches that improve patients' experiences and lower expenditures. This observational project assigned a lay health worker to conduct proactive symptom assessments intended to achieve these goals among patients with advanced cancer.

DETAILED DESCRIPTION:
All newly diagnosed Medicare Advantage enrollees with Stage 3 or 4 solid tumors or hematologic malignancies who planned to receive all oncology care at the Oncology Institute of Hope and Innovation from 11/1/2015 through 9/30/2016 were enrolled in the program. The program consisted of a 12-month telephonic program in which a lay health worker (LHW) supervised on-site by a registered nurse practitioner (RNP), assessed patient symptoms after diagnosis using the validated Edmonton Symptom Assessment Scale (ESAS) with the frequency of symptom assessment varying based on patient risk. We evaluated feasibility, defined as monthly LHW documentation of symptom assessments, and change in patient-reported satisfaction and overall and emotional and mental health with validated assessments at enrollment and 5-months post-enrollment among patients in the intervention. We compared healthcare use and costs to a historical cohort of similar Medicare Advantage enrollees diagnosed between 11/1/2014-10/31/2015 (control). We assessed differences in demographic and clinical factors between the two groups using chi-square and t-tests and used generalized linear models to evaluate differences in healthcare use and costs.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of stage 3 and 4 cancer
2. Clinical diagnosis of hematologic malignancy
3. Must receive care at the Oncology Institute of Hope and Innovation
4. Must be an enrollee of CareMore Medicare Advantage

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have a diagnosis of stage 3 and 4 cancers and who are receiving care at the Oncology Institute of Hope and Innovation and have CareMore Medicare Advantage as their healthcare payer plan.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was implemented with CareMore Health and the Oncology Institute of Hope and Innovation, which has 26 locations across southern California. Enrollment was conducted between November 1, 2015 and September 30, 2016. Each patient participated for 12 months or until death, whichever occurred first.
Pre-assignment Details: Patients were excluded from the intervention and control groups if they did not require medical oncology services.
Groups:
- Control Group: All participants in the control group received usual cancer care provided by Oncology Institute for Hope and Innovation clinics.
- Intervention Group: The intervention consisted of a 12-month telephonic program in which a lay health-worker (LHW), supervised by a physician assistant, assessed patient symptoms after diagnosis using the Edmonton Symptom Assessment Scale (ESAS) Participants were then sorted into two categories: High-risk or low-risk. For high-risk patients, the LHW conducted weekly telephone screenings until the patient's risk changed or death. For low-risk patients, the intervention was conducted by the LHW on a monthly basis.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 102 | 186
Completed | 100 | 183
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: All newly diagnosed Medicare Advantage enrollees with stage 3 or 4 solid tumors or hematologic malignancies who were receiving care in a community oncology practice.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 102 | 186 | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 102 | 186 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 (7.5) | 79 (8.0) | 79 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 101 | 158
  Male | 45 | 85 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity, No. (%): Non-Hispanic White | 49 | 88 | 137
  Race/Ethnicity, No. (%): Hispanic | 42 | 83 | 125
  Race/Ethnicity, No. (%): Non-Hispanic Black | 4 | 6 | 10
  Race/Ethnicity, No. (%): Asian Pacific Islander | 4 | 5 | 9
  Race/Ethnicity, No. (%): Native Hawaiian/Alaskan Native/American Indian | 3 | 4 | 7
Cancer Diagnosis [Count of Participants; unit: Participants]
  Thoracic | 13 | 29 | 42
  GI | 29 | 50 | 79
  Genitourinary | 15 | 33 | 48
  Malignant hematologic conditions | 14 | 18 | 32
  Breast | 18 | 23 | 41
  Other (i.e. skin, brain, bone, soft tissues, head/neck) | 13 | 33 | 46
Cancer Stage [Count of Participants; unit: Participants] — Cancer stages: stage 0 - the cancer is where it started (in situ) and hasn't spread; stage 1 - the cancer is small and hasn't spread anywhere else; stage 2 - the cancer has grown, but hasn't spread; stage 3 - the cancer is larger and may have spread to the surrounding tissues and/or the lymph nodes (or "glands", part of the immune system); stage 4 - the cancer has spread from where it started to at least 1 other body organ, also known as "secondary" or "metastatic" cancer. Stage was abstracted through chart review of clinical notes documented in the electronic health record by the oncologist.
  Participants
    3 | 47 | 71 | 118
    4 | 55 | 115 | 170

OUTCOME MEASURES:

1. Primary Outcome: Edmonton Symptom Assessment Scale Score (ESAS)
Description: ESAS measures participant responses to 10 common symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep problems, and feeling of well-being). Participants rate the intensity of 10 symptoms, each on a 11-point scale (0 to 10); sub-scores are then summed and averaged to create a total symptom score (range: 0 to 10, with 10 corresponding to worst symptom severity).
Time Frame: 12 months after patient enrollment
Population: Only participants in the intervention group were invited to complete the ESAS.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 0 | 186
score on a scale
  Symptom score at enrollment |  | 9.6 [0 to 10]
  Symptom score after 12 months |  | 7.2 [0 to 8]

2. Secondary Outcome: Incidence of Emergency Department Visits
Description: Emergency Department use for each patient abstracted from medical claims data review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Number; unit: visits per 1000 members/yr.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 102 | 186
visits per 1000 members/yr. | 0.92 | 0.61

3. Secondary Outcome: Hospitalization Visits (Claims Review)
Description: Hospitalization Use for each patient will be abstracted by medical claims data review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 102 | 186
number of visits
  No. of Admissions | 1.02 (1.44) | 0.72 (0.96)
  No. of readmissions | 0.10 (0.41) | 0.18 (0.47)

4. Secondary Outcome: Intensive Care Unit Visits (Claims Review)
Description: Intensive Care Unit Visits for each patient will be abstracted by medical claims data review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 102 | 186
number of visits | 0.66 (1.23) | 0.60 (1.00)

5. Secondary Outcome: Total Health Care Costs (Claims Review)
Description: Total Health Care Costs for each patient will be abstracted by medical claims data review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Median (Inter-Quartile Range); unit: $USD
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 102 | 186
$USD | 31,946 [15,754 to 57,369] | 21,266 [8,102 to 47,900]

6. Secondary Outcome: Change in Patient Satisfaction With Care Using the Consumer Assessment of Health Care Providers and Systems -General Survey
Description: Each patient will receive a satisfaction with care survey (The Consumer Assessment of Health Care Providers and Systems - General (CAHPS)) at baseline and 5 months. We will measure the change in satisfaction from calculated as the value at 5 months minus the baseline value. Scores for satisfaction were assessed using the Consumer Assessment of Healthcare Providers and Systems-General survey question #18 which measured rating of health provider, on which scores range from 0 to 10, with higher ratings correspond to higher patient satisfaction. Scores for each group are averaged at baseline and at 12 months.
Time Frame: Change in Patient Satisfaction with Care from baseline to 5 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 100 | 183
score on a scale
  Baseline (diagnosis) | 8.34 (1.83) | 8.10 (1.80)
  5-month follow-up | 8.10 (1.96) | 9.25 (1.03)
  Change at 5-months | -0.23 (1.88) | 1.15 (1.79)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between time of enrollment and 1 year
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 29/102 | 73/186
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/186
Other Adverse Events (participants affected / at risk) | 0/102 | 0/186

LIMITATIONS AND CAVEATS:
The study was limited to one community oncology practice and to a Medicare Advantage population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-03-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT03737058/Prot_000.pdf